CLINICAL TRIAL: NCT04214145
Title: The Effect of Phenylephrine, Norepinephrine and Vasopressin on Cerebral Oxygentaion During Off Pump CABG: A Pilot Study
Brief Title: The Effect of Vasopressors on Cerebral Oxygentaion During Off Pump CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPCAB_vasopressor
Record Dates: First submitted 2019-12-22; First posted 2020-01-02 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Oxygen Saturation
MeSH Terms: interventions — Phenylephrine; Norepinephrine; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phenylephrine (Experimental)
  Interventions: Drug: Phenylephrine
- Norepinephrine (Experimental)
  Interventions: Drug: Norepinephrine
- Vasopressin (Experimental)
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Phenylephrine — Continuous infusion of Phenylenphrine 250 μg/mL (=Phenylephrine 10mg * 5@ + D5W 200 mL) if mean BP < 60mmHg.
  1. Initial rate: 0.42 μg/kg/min (=0.1 mL/kg/hr)
  2. Increment by 0.21 μg/kg/min (=0.05 mL/kg/hr) if mean BP < 60mmHg after 5 minutes
  3. Maximum rate: 3.33 μg/kg/min (=0.8 mL/kg/hr)
  Arms: Phenylephrine
Drug: Norepinephrine — Continuous infusion of Norepienphrine 20 μg/mL (=NE 4mg * 1@ + D5W 200 mL) if mean BP < 60mmHg.
  1. Initial rate: 0.03 μg/kg/min (=0.1 mL/kg/hr)
  2. Increment by 0.015 μg/kg/min (=0.05 mL/kg/hr) if mean BP < 60mmHg after 5 minutes
  3. Maximum rate: 0.24 μg/kg/min (=0.8 mL/kg/hr)
  Arms: Norepinephrine
Drug: Vasopressin — Continuous infusion of Vasopressin 0.1 u/mL (=Vasopressin 20u * 1@ + D5W 200 mL) if mean BP < 60mmHg.
  1. Initial rate: 0.01 u/kg/hr (=0.1 mL/kg/hr)
  2. Increment by 0.005 u/kg/hr (=0.05 mL/kg/hr) if mean BP < 60mmHg after 5 minutes
  3. Maximum rate: 0.08 u/kg/hr (=0.8 mL/kg/hr)
  Arms: Vasopressin

SUMMARY:
The purpose of this study is to analyze the changes in cerebral oxygen saturation during the use of three vasopressors, phenylephrine, norepinephrine, and vasopressin, which are currently used during coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing off pump coronary artery bypass.

Exclusion Criteria:

* Patient refusal
* Preoperative vasopressor use
* Preoperative mechanical circulatory support
* Concurrent cerebrovascular or head and neck surgery
* Technical difficulty of measuring brain oxygen saturation
* Redo coronary artery bypass surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation (%) | during surgery
  continuous monitoring of cerebral oxygen saturation during surgery

SECONDARY OUTCOMES:
blood pressure | during surgery
  systolic/diastolic/mean blood pressure(mmHg)
heart rate | during surgery
  heart rate(/min)
cardiac index | during surgery
  cardiac index (L/min)
Total amount of infused drug | during surgery
  Propofol, remifentanil, vasoacitve drugs
Input/output | during surgery
  Urine output, blood loss, amount of fluid and transfusion
Sublingual microscopy | 1) After induction, 2) lateral wall or posterior wall anastomosis (if possible) 3) skin closure
  using SDF imaging device
Vascular occlusion test | 1) After induction, 2) lateral wall or posterior wall anastomosis (if possible) 3) skin closure
  using InspectraTM StO2
Troponin I | during surgery, at ICU admission, 24 hours / 48 hours after ICU admission
  Troponin I (ng/mL)
lactate | during surgery, at ICU admission, 24 hours / 48 hours after ICU admission
  lactate (mmol/L)
creatinine | during surgery, at ICU admission, 24 hours / 48 hours after ICU admission
  creatinine (mg/dL)
albumin | during surgery, at ICU admission, 24 hours / 48 hours after ICU admission
  albumin (g/dL)
NGAL | during surgery, at ICU admission, 24 hours / 48 hours after ICU admission
  NGAL (ng/mL)
MACCE | until 1 year after surgery
  Major adverse cardiac and cerebrovascular events
AKI/RRT | until 1 year after surgery
  renal complication

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul National University Hospital, Seoul, South Korea